CLINICAL TRIAL: NCT01190098
Title: Searching for "Sleep Friendly" Therapies for a Sleepy Population: A Double-Blind, Placebo-Controlled, Randomized Trial to Assess the Effects of Lacosamide on Sleep and Wake in Adults With Focal Epilepsy
Brief Title: Randomized Controlled Trial to Assess Effects of Lacosamide on Sleep and Wake in Adults With Focal Epilepsy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UCB-SLEEP
Record Dates: First submitted 2010-08-24; First posted 2010-08-27 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Partial Epilepsy
Keywords: Partial epilepsy; Excessive daytime sleepiness; Epworth Sleepiness Scale; Maintenance of Wakefulness Test
MeSH Terms: conditions — Epilepsies, Partial; Disorders of Excessive Somnolence | interventions — Lacosamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lacosamide (Experimental)
  Interventions: Drug: Lacosamide
- Sugar pill (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Lacosamide — Subjects randomized to lacosamide according to the following schedule:
  Treatment Phase Week Dose Week 1 LCM 50 mg bid Week 2 LCM 100 mg bid Week 3 LCM 150 mg bid Week 4 LCM 200 mg bid
  Other Names: LCM
  Arms: Lacosamide
Drug: Placebo — Placebo will be packaged identically to experimental drug and titrated according to the same schedule.
  Other Names: Control
  Arms: Sugar pill

SUMMARY:
Sleepiness and fatigue are the most common complaints of people with epilepsy and can have a negative impact on quality of life. Though unproven, these problems are often blamed on anti-seizure medications. The purpose of this study is to investigate the impact of the anti-seizure medication Lacosamide (Vimpat®) on sleep and wakefulness in adults with focal (partial onset) seizures.

Focal epilepsy, also called partial epilepsy, is a disorder characterized by seizures arising from a localized network of neurons in the brain. Focal seizures usually begin a sensation or involuntary movement of a part of the body, an unusual feeling, or a disturbance in hearing, smell, vision, or consciousness. The study is open to adults 18 and older with focal seizures.

Participation involves a physical exam, sleep testing at the Sleep Center, blood tests, completion of study questionnaires/diaries, and a random assignment to either take the study drug or placebo (often called a "look alike" or "sugar pill") for 5 to 8 weeks. There are 5 study visits. Participants will receive compensation for time spent in the study.

If you would like more information on this study please contact the Cleveland Clinic Sleep Center:

Dr. Nancy Foldvary-Schaefer: 216-445-2990 Monica Bruton: 216-444-6718

DETAILED DESCRIPTION:
1.1. Background Epilepsy is a common disorder affecting approximately 1% of the population including nearly 2 million people in the United States. Excessive daytime sleepiness (EDS) is the most common complaint of people with epilepsy, reported in as many 50% of cases. EDS has long been attributed to the effects of antiepileptic drugs (AEDs) and seizures, but this assumption has not been adequately tested. In recent years, primary sleep disorders, such as sleep apnea, have been identified as potential contributors. A recent questionnaire-based study of 486 adults with epilepsy found a 2-fold higher prevalence of sleep disturbances in patients compared with age- matched controls (39% vs.18%). The presence of a sleep disturbance adversely affects quality of life (QOL) in people with epilepsy.

Despite the frequency of EDS in people with epilepsy, surprisingly few have attempted to measure this complaint objectively. In a study presented at the 2007 Annual Meeting of the American Academy of Sleep Medicine (AASM) by the investigators of this proposal, the prevalence of EDS among 92 epilepsy patients was assessed using three measures: self-reported EDS, the Epworth Sleepiness Scale (ESS), a subjective screening tool used in sleep clinics, and the multiple sleep latency test (MSLT), the gold standard objective measurement of daytime sleepiness. Seventy-two percent of subjects endorsed EDS (feeling excessively sleepy at least a few days per week over the last 6 months), 37% had abnormal ESS scores (> 10), and 62% had abnormal MSLTs (mean sleep latency [MSL] < 8 min). The MSL was less than 5 minutes, comparable to that of patients with narcolepsy, in 36% of cases. The correlation between self-reported EDS and the MSL was poor. However, as found in previous studies in sleep populations, a better correlation between the ESS and MSL was found. Among larger epilepsy series using the ESS, 11-28% of patients had scores greater than 10, suggesting the presence of EDS.

Excessive daytime sleepiness is a negative predictor of QOL in sleep disorders patients and is likely the most important, overlooked complaint of people with epilepsy. To date, no well-designed trials have explored the impact of specific AED therapy on wakefulness, although the sedating effects of most of the currently available agents have been demonstrated through small series and clinical experience. The current study is proposed to objectively measure the effects of lacosamide (LCM) on sleep and wakefulness in adult patients with focal epilepsy.

1.2. Investigational Agent Lacosamide ([R]-2-acetamido-N-benzyl-3-methoxypropionamide) belongs to a novel class of functionalized amino acids. It has been shown in animal models to have antiepileptic properties possibly by two distinct and novel mechanisms of action. Like many other AEDs, LCM has an effect on voltage-gated sodium channels. But unlike other AEDs, LCM enhances the slow inactivation of these channels. LCM also interacts with collapsin-response mediator protein-2 (CRMP-2) which may represent other novel mechanism, not previously recognized in AED development.

Lacosamide 200-400 mg/day is approved in the US and in Europe in oral and IV formulations as adjunctive therapy in adults with focal seizures.

2.0 STUDY OBJECTIVES Primary Objective To determine the effect of LCM on wakefulness in adults with focal epilepsy by comparing the change between Visit 4 and baseline in the ESS in subjects randomized to LCM versus placebo.

Secondary Objectives

1. To determine the effect of LCM on wakefulness in adults with focal epilepsy by comparing the change between Visit 4 and baseline in MSL of the Maintenance of Wakefulness Test (MWT) in subjects randomized to LCM versus placebo.
2. To determine the impact of LCM on sleep using ambulatory polysomnography (PSG) by comparing sleep efficiency (SE; total sleep time/total recording time) between Visit 4 and baseline in subjects randomized to LCM versus placebo.
3. To compare change in fatigue using the Fatigue Severity Scale (FSS) between Visit 4 and baseline in subjects randomized to LCM versus placebo.
4. To compare change in health- and sleep-related QOL between Visit 4 and baseline in subjects randomized to LCM versus placebo.

3.0 STUDY DESIGN This is a Phase IV, randomized, single center trial of LCM in adult subjects with focal epilepsy. Subjects who meet the inclusion criteria and are taking stable doses of 1 or 2 marketed AEDs for at least 4 weeks will be randomized in a double-blind, 4:1 scheme to LCM 400 mg/day or placebo, respectively. At the end of the Treatment Phase, subjects will have the option to enter an Extension Phase whereby they will receive LCM titrated to 400 mg/day.

4.0 STUDY DRUG Subjects will be randomized to LCM or identically packaged placebo. A 1-step, back-titration of LCM 100 mg/day or placebo will be allowed in the case of an intolerable adverse event (AE) at the end of the Treatment Phase.

A blocked randomization scheme will be developed and used to allocate subjects to active treatment or placebo in a 4:1 ratio. Blocks will be of random size, not to exceed 10, and will ensure appropriate balance of treatment groups at the midpoint of enrollment and study completion.

5.0 STUDY PROCEDURES

5.1 Study Assessments

5.1.1 Sleep Apnea Scale of the Sleep Disorders Questionnaire (SA/SDQ) As part of the screening process, subjects will complete the SA/SDQ, a validated instrument that assesses the likelihood of having obstructive sleep apnea (OSA) based on variables including loud snoring, age, body mass index, tobacco use, and hypertension. In the original validation, cutoffs of 32 or higher for women and 36 or higher for men correlated well with having a diagnosis of OSA by PSG.

The following procedures (subjective assessments, blood sampling and sleep testing will be performed at baseline (Visit 2- 2 week window) and at Visits 3 (LCM 200 mg/day) and 4 (400 mg/day) at least 11 days but no longer than 21 days after the prior visit (at least 11 days after the previous dose adjustment so as to ensure a steady state).

5.1.2 Ambulatory PSG Overnight ambulatory PSG will be performed using the Sapphire PSG ™, Cleveland Medical Devices, Inc. The system records electroencephalography (EEG; F3/4, C3/4, O1/2), electro-oculography (EOG; E1, E2), chin electromyography (EMG; 3 channels), leg EMG (4 channels), thermister and pressure transducer, respiratory effort (RIP), snore, EKG, pulse oximetry, and body position. Remote PSG monitoring with video will be performed using DreamPort™, Cleveland Medical Devices, Inc.

5.1.3 Maintenance of Wakefulness Test (MWT) The MWT is a modification of the more popular MSLT, the gold standard objective measurement of daytime sleepiness. The MSLT is intended to measure physiological sleep tendency under standardized conditions. It is based on the premise that the degree of sleepiness is reflected by sleep latency. The MWT is intended to measure one's ability to maintain wakefulness under standardized, relatively sedentary conditions.

5.1.4 Subjective Sleep Assessments Epworth Sleepiness Scale (ESS): The ESS is a self-administered eight-item questionnaire that measures a subject's subjective daytime sleep propensity. Subjects are asked how likely they are to doze off or fall asleep in 8 specific situations such as watching television or riding a car (never, slight, moderate, high: 0-3), with total scores ranging from 0-24. It has high test-retest reliability and a high level of internal consistency. An ESS score greater than 10 is considered indicative of EDS.

Self-reported EDS is categorized as a response of Yes or No to the question: Have you been feeling excessively sleepy at least a few days per week over the last 2 weeks?

Fatigue Severity Scale (FSS): The FSS is a validated method for assessing fatigue. It is comprised of 9 items that are rated according to a Likert-type scale from 1 to 7, where 1 indicates no impairment and 7 indicates severe impairment. Responses to individual items are tallied to produce a total score.

5.1.5 Seizure and Sleep Log Subjects will record sleep and wake times and quantify and characterize seizures in logs developed for the trial. Mean daily seizure frequency, excluding auras, between Baseline and Visit 4 will be calculated.

5.1.6 Adverse Events Assessments Adverse Event Profile (AEP): The AEP is an epilepsy-specific, 19-item questionnaire designed to monitor the frequency of common AEs associated with AEDs. Subjects rate the frequency of problems or side effects on a scale from 1 (Never) to 4 (Always or often).

Patient Health Questionnaire (PHQ-9): The PHQ-9 is a 9-item depression scale based on the diagnostic criteria for major depressive disorders in the Diagnostic and Statistical Manual Fourth Edition (DSM-IV). It is used in the diagnosis of depression and monitoring of treatments impacting on depression. A score of 10 and higher is indicative of moderate to severe depression. The PHQ-9 discriminates well between individuals with and without depressive disorders.

5.1.7 Quality of Life Assessments Quality of Life in Epilepsy (QOLIE-31): The QOLIE-31 is a 31-item survey of health-related quality of life for adults with epilepsy. The survey is derived from a longer, 89-item instrument.

Pittsburgh Sleep Quality Inventory (PSQI): The PSQI is a self-rating questionnaire for measuring subjective sleep quality. A global score is produced that represents the sum of seven component scores, each which addresses a specific aspect of subjective sleep quality.

Functional Outcomes of Sleep Questionnaire (FOSQ): The FOSQ is a self-administered 30-item questionnaire that offers a measurement of functional status as it relates to the impact of daytime sleepiness on daily activities. It measures the effect on activity level, vigilance, intimacy and sexual relationships, general productivity and social outcome.

5.2 Subjects will have 5 or 6 visits Visit 1 (Baseline Phase - 2 weeks) Visit 2 (Randomization, Start of Treatment Phase - at least 2 weeks after Visit 1 not to exceed 8 weeks) Visit 3 (Treatment Phase, LCM 200 mg/day - 11 -21 days after Visit 2) Visit 4 (Treatment Phase, LCM 400 mg/day - 11-21 days after Visit 3)

At the completion of all study procedures, subjects will be offered the option of entering a 4-week Extension Phase or a 2-week Taper Phase. In the Extension Phase, the investigators and subjects will remain blinded to the initial group assignment but all subjects will be treated with LCM. Subjects in the LCM arm will continue on 400 mg/day. Those in the placebo arm will undergo a 4-week titration schedule. All subjects will continue to maintain a seizure and sleep diary.

Subjects who decline participation in the Extension Phase will undergo a 2-week Taper Phase whereby LCM will be tapered by 200 mg/day per week.

Visit 5 (Final Visit for Nonextenders, beginning of Extension Phase - 0-21 days after Visit 4) For subjects opting to enter the Extension Phase, subjective assessments only will be performed at least 4 days after initiation of LCM 200mg/day to ensure testing is completed after achieving a steady state.

Visit 6 (Extension Phase Final Visit - 26- 42 days after Visit 5)

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet the following inclusion criteria to be eligible for the study.

* Subject can provide written informed consent and is willing to comply with study procedures.
* Subject is at least 18 years of age.
* Subject has focal epilepsy with classifiable seizures according to the International Classification of Epileptic Seizures, 1981.11
* Subject is deemed to be an appropriate candidate for LCM adjunctive therapy.
* Subject has been maintained on a stable dose of 1 or 2 marketed AEDs for at least 4 weeks.

Exclusion Criteria:

Subjects must meet the following exclusion criteria to be eligible for the study.

* Subject has a history of a moderate or severe sleep apnea (apnea-hypopnea index [AHI] > 15), severe insomnia (habitual sleep duration < 4 hours) or narcolepsy.
* Subject has a score on the Sleep Apnea Scale of the Sleep Disorders Questionnaire (SA/SDQ) at screening of 32 or higher (female) and 36 or higher (male).
* Subject is currently participating or has participated within the last 2 months in a trial of an investigational drug or experimental device.
* Subject has seizures or seizures clusters that are not quantifiable.
* Subject has 6 or more seizures (excluding auras) in the 2-week Baseline Phase.
* Subject has a medical condition that could reasonably be expected to interfere with drug absorption, distribution, metabolism or excretion.
* Subject has any medical or psychiatric condition, which in the opinion of the investigator, could jeopardize the subject's health or would compromise the - Subject has a history of alcohol or drug abuse within the previous 2 years.
* Subject has an acute or sub-acutely progressive central nervous system disease.
* Subject is pregnant, breastfeeding or of childbearing age and not surgically sterile or practicing an acceptable form of contraception (barrier contraception, surgically sterilized, IUD, abstinence) for the duration of the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Foldvary-Schaefer, DO, Principal Investigator — Cleveland Clinic Neurological Institue
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 52 subjects randomized, 59 subjects enrolled. The 7 either were either screen failures or chose not to proceed with the study.
Period: Overall Study
Arm/Group | Lacosamide | Sugar Pill
Started | 42 | 10
Completed | 39 | 8
Not Completed | 3 | 2
Not completed — Adverse Event | 2 | 0
Not completed — Patient coomorbidity | 0 | 1
Not completed — Lack of transportation | 1 | 0
Not completed — Other | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lacosamide | Sugar Pill | Total
Number analyzed (Participants) | 42 | 10 | 52
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 10 | 51
  >=65 years | 1 | 0 | 1
Gender [Count of Participants; unit: Participants]
  Female | 29 | 7 | 36
  Male | 13 | 3 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 42 | 10 | 52
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 4 | 15
  White | 30 | 5 | 35
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 42 | 10 | 52

OUTCOME MEASURES:

1. Primary Outcome: Change in Epworth Sleepiness Scale Score From Baseline to Visit 4
Description: Scale 0 - 24 Higher scores indicate more severe symptoms
Time Frame: Baseline and Visit 4 (approximately 1 - 2 months)
Measure: Mean (95% Confidence Interval); unit: Units on a scale
Arm/Group | Lacosamide | Sugar Pill
Number analyzed (Participants) | 39 | 8
Units on a scale | -1.2 [-2.9 to 0.53] | -1.1 [-5.2 to 3.0]
Statistical Analysis 1: Comparison: Lacosamide vs Sugar Pill; Test type: Non-Inferiority or Equivalence — Null hypothesis: there is a non-inferiority region of 4 points; p = 0.027, t-test, 1 sided

2. Secondary Outcome: Change in the Fatigue Severity Scale From Baseline to Visit 4.
Description: Fatigue Severity Scale (FSS): Range 7- 63 where higher scores indicate more severe fatigue.
Time Frame: Baseline to Visit 4 (approximately 1 - 2 months)
Population: 6 subjects did not complete enough questions on the tool for the total score to be calculated at both time points.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lacosamide | Sugar Pill
Number analyzed (Participants) | 33 | 8
units on a scale | 0.30 [-3.7 to 4.3] | -5.4 [-17.1 to 6.4]
Statistical Analysis 1: Comparison: Lacosamide vs Sugar Pill; Test type: Superiority or Other; p = 0.23, t-test, 2 sided; Mean Difference (Net) = 5.7

3. Secondary Outcome: Change in Pittsburgh Sleep Quality Inventory (PSQI) From Baseline to Visit 4
Description: Range 0-21, where higher scores more impairment (in terms of sleep quality).
Time Frame: Baseline to Visit 4 (approximately 1 - 2 months)
Population: 7 subjects did not complete enough questions on the tool for the total score to be calculated at both time points.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lacosamide | Sugar Pill
Number analyzed (Participants) | 34 | 6
units on a scale | -1.6 [-2.9 to 0.0] | -1.3 [-2.9 to 0.3]
Statistical Analysis 1: Comparison: Lacosamide vs Sugar Pill; Test type: Superiority or Other; p = 0.84, t-test, 2 sided; Mean Difference (Net) = -0.3

4. Secondary Outcome: Change in Functional Outcomes of Sleep Questionnaire (FOSQ) From Baseline to Visit 4.
Description: Range 0-20 where lower scores indicate more impairment (sleep related QOL).
Time Frame: Baseline to visit 4 (approximately 1 - 2 months)
Population: 5 subjects did not complete enough questions on the tool for the total score to be calculated at both time points.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lacosamide | Sugar Pill
Number analyzed (Participants) | 34 | 8
units on a scale | 0.3 [0.0 to 1.0] | 1.1 [-1.3 to 3.5]
Statistical Analysis 1: Comparison: Lacosamide vs Sugar Pill; Test type: Superiority or Other; p = 0.37, t-test, 2 sided; Mean Difference (Net) = -0.8

5. Secondary Outcome: Change in Adverse Event Profile (AEP) From Baseline to Visit 4.
Description: Range 19-76, where higher scores indicate more severe impairment (in terms of 19 common antiepileptic drug side effects.
Time Frame: Baseline to visit 4 (approximately 1 - 2 months)
Population: 3 subjects did not complete enough questions on the tool for the total score to be calculated at both time points.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lacosamide | Sugar Pill
Number analyzed (Participants) | 37 | 7
units on a scale | -1.2 [-5.2 to 2.9] | -6.0 [-14.2 to 2.2]
Statistical Analysis 1: Comparison: Lacosamide vs Sugar Pill; Test type: Superiority or Other; p = 0.33, t-test, 2 sided; Mean Difference (Net) = 4.8

6. Secondary Outcome: Change in Patient Health Questionnaire-9 (PHQ-9) From Baseline to Visit 4.
Description: Range 0-27, where higher scores indicate more impairment (depressive symptoms)
Time Frame: Baseline to visit 4 (approximately 1 - 2 months)
Population: 5 subjects did not complete enough questions on the tool for the total score to be calculated at both time points.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lacosamide | Sugar Pill
Number analyzed (Participants) | 34 | 8
units on a scale | -1.1 [-2.7 to 0.6] | -1.2 [-4.6 to 2.1]
Statistical Analysis 1: Comparison: Lacosamide vs Sugar Pill; Test type: Superiority or Other; p = 0.92, t-test, 2 sided; Mean Difference (Net) = 0.1

7. Secondary Outcome: Change in Daily Seizure Frequency From Baseline to Visit 4
Description: Number of seizures per day.
Time Frame: Baseline to visit 4 (approximately 1 - 2 months)
Population: 2 subjects did not complete seizure diary at both time points.
Measure: Median (Inter-Quartile Range); unit: number of seizures per day
Arm/Group | Lacosamide | Sugar Pill
Number analyzed (Participants) | 37 | 8
number of seizures per day | 0.0 [0.0 to 0.15] | 0.0 [0.0 to 0.04]
Statistical Analysis 1: Comparison: Lacosamide vs Sugar Pill; Test type: Superiority or Other; p = 0.69, Wilcoxon (Mann-Whitney); Median Difference (Net) = 0.0

8. Secondary Outcome: Change in Quality of Life in Epilepsy (QOLIE-31) From Baseline to Visit 4
Description: Range 0 -10 where higher scores reflect better quality of life.
Time Frame: Baseline to visit 4 (approximately 1 - 2 months)
Population: 5 subjects did not complete enough questions on the tool for the total score to be calculated at both time points.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Lacosamide | Sugar Pill
Number analyzed (Participants) | 36 | 6
units on a scale | 4.0 [1.2 to 6.7] | 4.2 [-2.3 to 10.6]
Statistical Analysis 1: Comparison: Lacosamide vs Sugar Pill; Test type: Superiority or Other; p = 0.95, t-test, 2 sided; Mean Difference (Net) = -0.2

ADVERSE EVENTS:
Time Frame: Visit 2 - Visit 4, approximately 1 to 2 months.
Arm/Group | Lacosamide | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 3/42 | 0/10
Other Adverse Events (participants affected / at risk) | 37/42 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lacosamide (N=42) | Sugar Pill (N=10)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Increased seizures (Nervous system disorders) | 1 (1) | 0 (0)
Accidental overdose (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Lacosamide (N=42) | Sugar Pill (N=10)
Heart palpitations (Cardiac disorders) | 1 | 2
Common cold/flu (Immune system disorders) | 9 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Infection (Infections and infestations) | 1 | 1
Skin burn/abrasion/bruise (Injury, poisoning and procedural complications) | 3 | 0
Ataxia (Nervous system disorders) | 4 | 1
Blurred vision (Nervous system disorders) | 8 | 1
Diplopia (Nervous system disorders) | 3 | 0
Shaky hands (Nervous system disorders) | 3 | 0
Fall with injury (Injury, poisoning and procedural complications) | 2 | 1
Dizziness (Nervous system disorders) | 18 | 3
Fatigue (Nervous system disorders) | 4 | 2
Headache (Nervous system disorders) | 17 | 4
Memory impairment (Nervous system disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 7 | 2
Somnolence (Nervous system disorders) | 3 | 0
Tremor (Nervous system disorders) | 4 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No